CLINICAL TRIAL: NCT01007747
Title: EPT 100: Geranium Oil for the Relief of Neuropathic Pain
Acronym: Geranium Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 21033
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Neuropathic Pain
Keywords: Geranium oil; Neuropathy
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Geranium oil (Experimental)
  Interventions: Other: Geranium oil

INTERVENTIONS:
Other: Geranium oil — Daily topical application over neuropathic pain

SUMMARY:
The purpose of this study is to determine if Geranium oil will relieve a variety of neuropathic pain and some pain relief will last more than 48 hours.

DETAILED DESCRIPTION:
EPT 100 study is designed to identify the percentage of people who experience neuropathic pain relief from topical geranium oil from Reunion Island, determine which neuropathic pain conditions respond best and define the time course of the pain relief.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or oler
* Neuralgia or neuropathy with daily pain
* At least moderate intensity pain
* Signed informed consent

Exclusion Criteria:

* Pregnant or nursing
* Known allergies to geranium oil or geranium oil fractions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain relief | 3 times in 30 to 60 minutes post-application

SECONDARY OUTCOMES:
Response to therapy at 30 to 60 minutes, they will be asked to apply the oil to painful area daily | Daily over 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States